CLINICAL TRIAL: NCT05822479
Title: Bilateral Ultrasound-guided External Oblique Intercostal Block for Postoperative Analgesia in Patients Undergoing Laparoscopic Sleeve Gastrectomy Surgery: A Prospective Randomized Controlled Study
Brief Title: Laparoscopic Sleeve Gastrectomy Surgery and External Oblique Intercostal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Cengiz KAYA, Principal Investigator, Clinical Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: EOIB2022
Record Dates: First submitted 2023-04-10; First posted 2023-04-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia; Regional Anesthesia; Morbid Obesity; Postoperative Pain
Keywords: Anesthesia; Nerve block; Obesity; Laparoscopy; External oblique intercostal block
MeSH Terms: conditions — Obesity, Morbid; Pain, Postoperative; Obesity

STUDY DESIGN:
Intervention Model Description: A block randomization list will be created by a doctor who does not participate in patient follow-up using a web-based program, 'Research Randomizer (Urbaniak and Plous, 2013)'.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed opaque envelopes containing study participation numbers will be used to assign each patient. A researcher not involved in patient follow-up will use the web-based "Research Randomizer" (Urbaniak and Plous 2013) tool to give each participation number to a random group with a 1:1 ratio. A nurse not an active investigator in the study will have each participant choose an envelope containing the study participation number. They will inform the anesthetist administering the block/blocks about which group the patient is in immediately before administration. Researchers, surgeons, and nurses will not be aware of the randomization of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group EOIB (Active Comparator): A bilateral EOIB (60 ml, %0.25 bupivacaine, totally) + IV morphine patient-controlled analgesia (PCA)
  Interventions: Procedure: Bilateral ultrasound guided external oblique intercostal block (EOIB)
- Group Control (Other): IV morphine PCA
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Bilateral ultrasound guided external oblique intercostal block (EOIB) — Bilateral ultrasound-guided EOIB (total of 60 ml, %0.25 bupivacaine) will be performed + IV morphine PCA
  Multimodal analgesia :
  Patients are administered iv tenoxicam 20mg and tramadol 100 mg after induction of general anesthesia, iv paracetamol 1 gr and iv morphine 0.05 mg/kg/ideal body weight (IBW) will be administered. Postoperative analgesia: iv paracetamol 1gr every 8 hours and IV PCA of 0,5mg/ml morphine (the bolus dose is 20 µg/kg, the lock-in time of 10 minutes, the 4-hour limit is adjusted to be 80% of the calculated total amount). Rescue analgesia, when necessary (if the resting NRS score is ≥4 despite PCA demand), 25 mg IV meperidine was administered in the recovery unit, and 50 mg intramuscular (IM) meperidine was administered in the ward.
  Other Names: External oblique intercostal block
  Arms: Group EOIB
Other: Control — Patients in this group will not be performed interfacial plane blocks.
  Multimodal analgesia :
  Patients are administered iv tenoxicam 20mg and tramadol 100 mg after induction of general anesthesia, iv paracetamol 1 gr and iv morphine 0.05 mg/kg/ideal body weight (IBW) will be administered. Postoperative analgesia: iv paracetamol 1gr every 8 hours and IV PCA of 0,5mg/ml morphine (the bolus dose is 20 µg/kg, the lock-in time of 10 minutes, the 4-hour limit is adjusted to be 80% of the calculated total amount). Rescue analgesia, when necessary (if the resting NRS score is ≥4 despite PCA demand), 25 mg IV meperidine was administered in the recovery unit, and 50 mg IM meperidine was administered in the ward.
  Arms: Group Control

SUMMARY:
In obese patients, adequate pain relief in the postoperative period is an important parameter that affects patient comfort and hospital stay. Increasing patient comfort and recovery quality can be achieved by avoiding undesirable effects such as nausea, vomiting, and analgesia. This study aimed to evaluate the impact of the external oblique intercostal block postoperative acute pain scores and opioid consumption in the first 24 hours after laparoscopic sleeve gastrectomy surgery.

DETAILED DESCRIPTION:
Adequate pain control in laparoscopic surgeries is associated with reduced postoperative opioid administration, faster mobilization, faster recovery, and shorter hospital stays. Intraoperative nerve blocks using local anesthetics have been shown to improve postoperative pain in various abdominal surgeries, both open and laparoscopic. Laparoscopic bariatric procedures are most often associated with moderate to severe visceral pain from surgical manipulation of the stomach and intestine. Combined regional and general anesthesia reduces surgical stress responses by interrupting pain transmission signals, which facilitates pain control, reduces opioid consumption, and improves patient postoperative satisfaction. Ultrasound-guided fascial plane blocks have been rapidly included in regional anesthesia applications as an alternative to neuraxial techniques in recent years and include injection into a tissue plane to provide analgesia in various anatomical areas. The external oblique intercostal block (EOIB) represents an essential modification of the fascial plane block techniques that can consistently cover the upper lateral abdominal wall. The EOIB block has easily identifiable sonographic points.

The study aims to investigate the effects of the EOIB on postoperative pain in morbidly obese patients who will undergo laparoscopic sleeve gastrectomy by comparing it with the control group. It is seen that there are not enough studies on EOIB in the literature. Our study, which the investigators think will contribute to the literature, was planned as a prospective, randomized, controlled, single-blind, parallel-group study.

Patients will be divided into two groups:

Group EOIB :

A bilateral EOIB (60 ml 0.25% bupivacaine + 1:400.000 adrenaline) will be performed. In addition, IV morphine-PCA will be applied postoperatively for 24 hours.

Group Control:

Patients in this group will not receive any block. IV morphine-PCA will be applied postoperatively for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Age between18-65 years
2. American Society of Anesthesiology score II-III
3. Body mass index (BMI) > 35 kg/m2
4. Patients who will sign the informed consent form

Exclusion Criteria:

1. Patients with drug allergies (Opioids, NSAIDs, local anesthetics)
2. Patients with neuro-psychiatric disease, cognitive impairment, inability to communicate, or a history of drug addiction
3. Presence of any systemic infection or at the injection site
4. Patients taking anticoagulants or having any bleeding disorder (Coagulopathy, International Normalized Ratio (INR) value not within normal limits, thrombocytopenia or platelet dysfunction)
5. Patients with significant cardiovascular, hepatic, renal or endocrine disorders
6. Patients with a history of chronic pain syndromes or receiving chronic pain treatment and a history of opioid use for more than four weeks in the preoperative period
7. Patients using continuous positive airway pressure device due to obstructive sleep apnea syndrome (OSAS) (symptoms detected by polysomnography and apnea-hypopnea index (AHI) >5/hour)
8. Patients with chronic obstructive pulmonary disease
9. Patients who need intensive care unit after surgery
10. Patients who do not consent/do not want to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption in the first 24 hours after surgery | postoperative day 1
  Cumulative opioid consumption in the first 24 hours after surgery will be measured. Patients can request opioids via a PCA device when their NRS score is ≥4. In cases where rescue analgesia is required (NRS score ≥4), 25 mg IV meperidine was administered in the recovery unit, and 50 mg IM meperidine was administered in the ward.

SECONDARY OUTCOMES:
Cumulative opioid consumption in the first 12 hours after surgery | postoperative day 1
  Cumulative opioid consumption in the first 12 hours after surgery will be measured. Patients can request opioids via a PCA device when their NRS score is ≥4 and 25 mg IV meperidine was administered in the recovery unit, and 50 mg IM meperidine was administered in the ward.
Postoperative pain scores | postoperative day 1
  Pain status at rest and while activity will be assessed by NRS score at 0, 3, 6, 12, 18, and 24 hours after surgery. The NRS is an 11-point numeric scale that ranges from 0 to 10.
Patients' satisfaction and quality of pain management | postoperative day 1
  Patients' pain management satisfaction and quality will be evaluated using the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) -Turkish Version.
The scores of postoperative nausea and vomiting (PONV) and the number of patients requiring postoperative antiemetics. | postoperative day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, 18, and 24 hours after extubation. For PONV prophylaxis, patients will be routinely administered 8 mg IV dexamethasone before induction and 0.15 mg/kg (IVA) IV ondansetron 20 minutes before the end of the procedure. If a score of 3 or more is recorded, 4 mg IV ondansetron will be administered and repeated after 4 hours if required. Despite the administration of ondansetron, if the score is ≥3, the patients will be administered 10 mg IV metoclopramide diluted in 100 ml saline solution as an IV infusion. The number of patients who receive antiemetic treatment will be recorded. The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once.
The number of patients who required rescue analgesia. | postoperative day 1
  The number of patients requiring rescue analgesics will be recorded over 24 hours.
Time of first analgesic request | postoperative day 1
  Time at which the first analgesic is requested
Intraoperative remifentanil consumption | The remifentanil consumption will be recorded from anesthesia induction until the patient is referred to the recovery unit, up to 150 minutes.
  The total amount of remifentanil consumed will be recorded.
The number of patients with complications | Postoperative 7 days on an average
  The number of patients has any complications -directly related to the block or the drug used in the block- will be recorded
The heart rate measurement | The heart rate was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit, up to 180 minutes.
  The heart rate was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit.
The mean arterial pressure measurement | The mean arterial pressure was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit, up to 180 minutes.
  The mean arterial pressure was recorded preoperatively, one minute after the induction, and every 15-30 minutes until the patient was referred to the recovery unit.

CONTACTS AND LOCATIONS:
Overall Officials: Cengiz KAYA, Study Director — Ondokuz Mayıs University Faculty of Medicine
Locations (1):
- Ondokuz Mayis Universitesi, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saber AA, Lee YC, Chandrasekaran A, Olivia N, Asarian A, Al-Ayoubi S, DiGregorio R. Efficacy of transversus abdominis plane (TAP) block in pain management after laparoscopic sleeve gastrectomy (LSG): A double-blind randomized controlled trial. Am J Surg. 2019 Jan;217(1):126-132. doi: 10.1016/j.amjsurg.2018.07.010. Epub 2018 Aug 1. PMID 30170687
- [Background] Elsharkawy H, Kolli S, Soliman LM, Seif J, Drake RL, Mariano ER, El-Boghdadly K. The External Oblique Intercostal Block: Anatomic Evaluation and Case Series. Pain Med. 2021 Nov 26;22(11):2436-2442. doi: 10.1093/pm/pnab296. PMID 34626112
- [Background] White L, Ji A. External oblique intercostal plane block for upper abdominal surgery: use in obese patients. Br J Anaesth. 2022 May;128(5):e295-e297. doi: 10.1016/j.bja.2022.02.011. Epub 2022 Mar 3. No abstract available. PMID 35249704
- [Background] Coskun M, Yardimci S, Arslantas MK, Altun GT, Uprak TK, Kara YB, Cingi A. Subcostal Transversus Abdominis Plane Block for Laparoscopic Sleeve Gastrectomy, Is It Worth the Time? Obes Surg. 2019 Oct;29(10):3188-3194. doi: 10.1007/s11695-019-03984-4. PMID 31175560